CLINICAL TRIAL: NCT02357186
Title: Multicenter Prospective Broad Validation of a Management Algorithm Mild Head Injury in Children
Brief Title: Broad Validation Study of a Management Algorithm Mild Head Injury in Children
Acronym: EVEACE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0038
Record Dates: First submitted 2015-01-21; First posted 2015-02-06 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Head Injury
Keywords: Mild head injury - clinical decision rule - Child
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Head injury is a frequent reason for consultation with pediatric emergencies, over 95% are mild head injury defined by a Glasgow score greater than or equal to 13. In October 2009, the Pediatric Emergency Care Applied Research Network has published a rule clinical decision support of mild head injury of the child with the aim to identify children at very low risk for clinically severe intracranial lesions in order to avoid the use of CT and unnecessary exposure to radiation ionizing. This clinical decision rule constructed from a multicenter prospective cohort 42,412 American children allows on anamnestic and clinical elements to guide medical decision for conducting brain imaging, hospital monitoring or discharge home placing the child in three levels of risk of clinically severe intracranial lesions.

Since March 2012, the French Emergency Medicine Society recommends for the treatment of mild head trauma the child's use of the clinical decision rule provided that it is the subject of a validation study externally. Indeed, after the construction phase and before its daily application, a clinical decision rule must be subject to an broad validation process so that its predictive performance can be definitively established.

The investigators' work aims to conduct this broad validation study prospective multicenter way in a French pediatric population, as recommended by the French Emergency Medicine Society, in order to confirm or deny its predictive performance and allow its application and generalization. The investigators will check and if the Rule Clinical Decision is adapted or not to the management of mild head injuries in the French pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children under 16 years admitted to an emergency room for mild head injury (Glasgow Coma Scale score ≥14) in the previous 24 hours
* Children who have agreed to participate in the study (if age> 8 years)
* Patient Parents have accepted the participation of their child in the study

Exclusion Criteria:

* Children with bleeding disorders
* Ventricular shunt Presence
* Benin mechanism of trauma (fall of the height of the child or impact against an object while walking / running with no sign that the scalp dermabrasion)
* Penetrating trauma
* Known brain tumor
* Previously known neurological disorders
* Evaluation scanographic in another hospital before emergency review

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Will be included in the study all children under 16 years of age admitted to the emergency room with mild head trauma with a Glasgow score greater than or equal to 14, occurred in the previous 24 hours. The mild head injury is usually defined by a GCS ≥ 13, but the study of the Pediatric Emergency Care Applied Research Network was interested in the population of children with TBI Glasgow score was greater than or equal to 14. Indeed the care of children with head trauma with a Glasgow score below 14 is not controversial. The risk of traumatic brain injury is at least 20%, achieving a brain scan is routinely recommended for these children. The investigators will resume the same characteristics for the study population as the study of the Pediatric Emergency Care Applied Research Network.
Sampling Method: Non-Probability Sample
Enrollment: 7871 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically severe intracranial injury and classified at risk (top and middle) according to clinical decision rule in all patients with severe intracranial lesions. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Fleur Lorton, Dr, Principal Investigator — Nantes University Hospital
Locations (9):
- France (9):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Centre Hospiatlier Départemental de Vendée, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Saint-Nazaire Hospital, Saint-Nazaire
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours